CLINICAL TRIAL: NCT05355779
Title: Needs Assessment to Guide the Development of a Paediatric Survivorship Programme in Hong Kong to Promote Physical and Psychological Well-being of Children After Cancer Treatment
Brief Title: Needs Assessment to Guide the Development of a Paediatric Survivorship Programme in Hong Kong
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Other Study IDs: HKCH-REC-2021-056
Record Dates: First submitted 2022-01-24; First posted 2022-05-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Cancer; Survivorship
Keywords: Paediatric Cancer; Survivorship; Post-treatment; Transition period; Qualitative study; Rehabilitation; Needs; Preferences
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interviewees: Paediatric cancer survivors, their parent/caregiver and health care professionals will be invited to express their views and perspectives in an interview with the researcher
  Interventions: Other: Not Application as this is a qualitative study

INTERVENTIONS:
Other: Not Application as this is a qualitative study — Not Application as this is a qualitative study

SUMMARY:
This study aims to fill the gaps in knowledge regarding the effects of cancer and its treatment on Hong Kong Chinese paediatric cancer survivors, especially during the transition period, to further capture a deeper understanding of the challenges, views and needs of Hong Kong Chinese paediatric cancer survivors and the key stakeholders around them via face-to-face conversations.

DETAILED DESCRIPTION:
Objectives: Although increasing attention has been devoted to the development of paediatric cancer survivorship programmes, most of these studies have originated in Western countries. Given the cultural differences between Asian and Western communities, the applicability of the findings to paediatric cancer survivors in Asian cultural contexts is limited. To date, research remains scant regarding the needs and challenges of Hong Kong Chinese paediatric cancer survivors and the key stakeholders involved during the transition period after cancer treatment. Although Hong Kong paediatric cancer survivors do attend regular medical follow-up visits, most attention has been focused on their physiological care, while their psychosocial needs remain unmet. Accordingly, the aim of this proposed study will be to fill the gaps in knowledge regarding the effects of cancer and its treatment, especially will focus on psychosocial effects in Hong Kong Chinese paediatric cancer survivors during the transition period.

Design and subjects: A qualitative descriptive design will be used. A purposive sample of 15 paediatric cancer survivor participants and their parents or caregivers, five paediatric oncology nurses and three paediatric oncologists will be invited for a semi-structured interview conducted with the aid of an interview guide.

Data analysis: A thematic analysis approach will be used for data analysis.

Expected results: The findings of this study will provide an in-depth understanding of the needs, challenges and views of paediatric cancer survivors and other key stakeholders, which will greatly facilitate the future development of appropriate targeted paediatric cancer survivorship programmes.

ELIGIBILITY:
Inclusion Criteria:

* able to speak Cantonese and read Chinese
* aged between 9 and 18 years of age
* Should have completed cancer treatment between 2 months and 2 years earlier

Exclusion Criteria:

* Children who received a diagnosis and completed treatment before the age of 9 will be excluded as they might have vague memories of the course of cancer and may have limited verbal and cognitive ability to express themselves
* Children of exclude parents will be exclueded

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric cancer survivors
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
An individual, a face-to-face interview will be conducted with the participants to identify the needs of paediatric cancer survivors during the transition period after cancer treatment | through study completion, an average of 15 months
  Semi-structured and open-ended questions will be used to collect qualitative data from the participants
An individual, a face-to-face interview will be conducted with the participants to assess the key elements in the development of a paediatric survivorship programme | through study completion, an average of 15 months
  Semi-structured and open-ended questions will be used to collect qualitative data from the participants

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chung, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Children's Hospital, Hong Kong, Hong Kong